CLINICAL TRIAL: NCT00191841
Title: Gemcitabine Plus Cisplatin as Neoadjuvant Chemotherapy in Operable Non Small Cell Lung Cancer
Brief Title: Gemcitabine in Combination With Cisplatin as Neoadjuvant NSCLC Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7410; B9E-VI-S327
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-07-24 (Estimated); Status verified 2006-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin

INTERVENTIONS:
Drug: gemcitabine
Drug: Cisplatin

SUMMARY:
To evaluate the clinical response rate of neoadjuvant chemotherapy with gemcitabine and cisplatin in patients with operable NSCLC

ELIGIBILITY:
Inclusion Criteria:

* histologic or cytologic diagnosis of operable non-small cell lung cancer (IB-IIIA)
* no prior chemotherapy
* WHO criteria for disease status assessment

Exclusion Criteria:

* Concurrent administration of any other tumor therapy
* pregnant or breast feeding
* serious concomitant disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-12; Study Completion 2006-02

PRIMARY OUTCOMES:
Antitumor activity

SECONDARY OUTCOMES:
Duration of response, time to progressive disease, time to treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Barnaul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ufa

REFERENCES:
- [Derived] Davidov MI, Polotzky BE, Marenich AF, Orlov SV, Lazarev AF, Skryabina LS, Pavlushkov EV, Semenchenya VA, Brichkova OY, Karaseva VV. Gemcitabine combined with cisplatin as neoadjuvant chemotherapy in stage IB-IIIA non-small cell lung cancer. Anticancer Drugs. 2011 Jul;22(6):569-75. doi: 10.1097/CAD.0b013e328342d50a. PMID 21487288